CLINICAL TRIAL: NCT01593124
Title: Identification of Novel Biomarkers of Cervicovaginal Mucosal Inflammation
Acronym: Biomarkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D11-119
Record Dates: First submitted 2012-03-09; First posted 2012-05-07 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Vaginal Inflammation; Vaginal Infections
Keywords: Vaginal innate immune and inflammatory responses
MeSH Terms: conditions — Vaginitis | interventions — Imiquimod; hydroxyethylcellulose; Nonoxynol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Imiquimod, 2 doses, vaginally (Active Comparator): Participants first have sampling in the follicular and luteal phases of the menstrual cycle. Then participants receive 4 doses of HEC placebo gel in the luteal phase. Finally, participants are randomized to the order of IMiquimod, 2 doses vaginally, in the luteal phase and nonoxynol-9, 4%, 4 doses vaginally in the luteal phase.
  Interventions: Drug: Imiquimod
- Placebo (Placebo Comparator): Participants first have sampling in the follicular and luteal phases of the menstrual cycle. Then participants receive 4 doses of HEC placebo gel in the luteal phase. Finally, participants are randomized to the order of IMiquimod, 2 doses vaginally, in the luteal phase and nonoxynol-9, 4%, 4 doses vaginally in the luteal phase.
  Interventions: Other: Placebo
- Nonoxynol-9 (Active Comparator): Participants first have sampling in the follicular and luteal phases of the menstrual cycle. Then participants receive 4 doses of HEC placebo gel in the luteal phase. Finally, participants are randomized to the order of IMiquimod, 2 doses vaginally, in the luteal phase and nonoxynol-9, 4%, 4 doses vaginally in the luteal phase.
  Interventions: Drug: Nonoxynol-9

INTERVENTIONS:
Drug: Imiquimod — Participants first have sampling in the follicular and luteal phases of the menstrual cycle. Then participants receive 4 doses of HEC placebo gel in the luteal phase. Finally, participants are randomized to the order of IMiquimod, 2 doses vaginally, in the luteal phase and nonoxynol-9, 4%, 4 doses vaginally in the luteal phase.
  Other Names: Aldara
  Arms: Imiquimod, 2 doses, vaginally
Other: Placebo — Participants first have sampling in the follicular and luteal phases of the menstrual cycle. Then participants receive 4 doses of HEC placebo gel in the luteal phase. Finally, participants are randomized to the order of IMiquimod, 2 doses vaginally, in the luteal phase and nonoxynol-9, 4%, 4 doses vaginally in the luteal phase.
  Other Names: Hydroxyethylcellulose
  Arms: Placebo
Drug: Nonoxynol-9 — Participants first have sampling in the follicular and luteal phases of the menstrual cycle. Then participants receive 4 doses of HEC placebo gel in the luteal phase. Finally, participants are randomized to the order of IMiquimod, 2 doses vaginally, in the luteal phase and nonoxynol-9, 4%, 4 doses vaginally in the luteal phase.
  Other Names: Conceptrol
  Arms: Nonoxynol-9

SUMMARY:
This study investigates the response of vaginal and cervical tissue after exposure to three vaginal products: hydroxyethyl cellulose (HEC) placebo, nonoxynol-9 (N9) and imiquimod (IMQ) cream.

DETAILED DESCRIPTION:
Each woman in this study will be evaluated 5 separate times:

1. Baseline in the follicular phase of the menstrual cycle;
2. Baseline in the luteal phase of the menstrual cycle;
3. After a 3 day (4 dose) treatment with HEC placebo;
4. After a 3 day (4 dose) treatment of 4% N-9;
5. After a 2 day (2 dose) treatment of IMQ.

A subset of 5 women will have an additional baseline visit in the follicular phase.

The order of the N-9 and IMQ treatments is randomized. The study is cross over in design. The per sequence of treatments is as follows: Baseline in the follicular phase of the menstrual cycle, next is baseline in the luteal phase of the menstrual cycle, next is after a 3 day (4 dose) treatment with HEC placebo. At this point in the study, half of the participants are randomized to do the N-9 treatment and then the IMQ treatment. The remaining half of the participants do the IMQ treatment and then the N-9 treatment.

All participants are sampled at the 5 timepoints described above.

ELIGIBILITY:
Inclusion Criteria:

1. 21 to 45 years of age, inclusive;
2. In good health, as evidenced by history and procedures at screening and enrollment visits without any clinically significant systemic disease;
3. Not be at risk for pregnancy, due to surgical sterilization of participant and or her sexual partner, abstinence for duration of study, consistent condom use, non-hormonal IUD or same sex relationship. Note: If consistent condom user, must agree to use condoms without spermicide for duration of study.;
4. Have had regular menstrual cycles (every 24-35 days) for the past two cycles;
5. Willing and able to comply with study procedures

Exclusion Criteria:

1. A clinically significant history of an abnormal pap smear (by written report) that has not been evaluated and or treated, if indicated, according to standard guidelines;
2. It has been less than 9 months since the participant's last depot medroxyprogesterone acetate (DMPA) injection and she has not had 2 normal, spontaneous menses (this can be shortened to 6 months if the participant has had at least 2 normal spontaneous menses);
3. Use of any other hormonal contraceptive method within past 3 months (oral, transdermal, transvaginal, implant, or intrauterine device) without 2 subsequent, normal menses;
4. Surgery or biopsy of the vulva, vagina, or cervix (including piercings) within 30 days;
5. Pregnancy within the past 3 months;
6. Currently breastfeeding;
7. Current STI or lower genital tract infection (including, but not limited to HIV-1, HSV-2, Chlamydia trachomatis (CT), Trichomonas vaginalis (TV), Neisseria Protocol # D11-119 Version 2.0 April 13, 2012 10 gonorrhea (NG), Hepatitis B, high risk HPV sub types and or Syphilis), yeast vaginitis or bacterial vaginosis (BV);
8. Current use of chronic immunosuppressants (for example daily steroids or daily non-steroidal anti-inflammatory drugs [NSAIDs]);
9. Current presence of vulvar, anal and or vaginal genital warts;
10. Current tobacco use of any amount;
11. Other conditions that, in the opinion of the investigator, would constitute contraindications to participation in the study or would compromise the ability to comply with study protocols, such as any major chronic illness including but not limited to cancer, serious autoimmune disease, metabolic disorders or a major psychiatric disorder (e.g., schizophrenia); and
12. Current participation in any other drug or device study, or any study which, in the

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Differential Microarray gene expression (particularly looking at pathways involved in inflammation and immune response) in vaginal tissues after exposure to N9, HEC or imiquimod | Biopsies are performed 8 - 18 hours after exposure to each product
  These data are still undergoing analysis

CONTACTS AND LOCATIONS:
Overall Officials: Andrea R Thurman, MD, Principal Investigator — CONRAD Clinical Research Center, Eastern VA Medical School
Locations (1):
- Eastern Virginia Medical School CONRAD Clinical Research Center, Norfolk, Virginia, United States

REFERENCES:
- See also: Study Sponsor — http://conrad.org